CLINICAL TRIAL: NCT00599053
Title: Early Versus Expectant Treatment of Ureaplasma Infection in Very Low Birth Weight Neonates
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment was terminated early due to a change in practice on the obstetrical side that included administering azithromycin to women with preterm labor.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert Schelonka, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F061228003
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Bacteria Infection; Respiratory Tract Infections
Keywords: Ureaplasma; Bronchopulmonary dysplasia; very low birthweight
MeSH Terms: conditions — Respiratory Tract Infections; Bronchopulmonary Dysplasia | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early treatment with azithromycin
  Interventions: Drug: Azithromycin
- 2 (No Intervention): Expectant (usual) management

INTERVENTIONS:
Drug: Azithromycin — 10 mg/kg IV per dose given for 10 days
  Arms: 1

SUMMARY:
Our hypothesis is that treatment of known Ureaplasma spp. infection of the airways in very low birth weight (VLBW) infants with azithromycin will eradicate the organisms and lessen the proinflammatory state caused by infection that puts them at risk for Bronchopulmonary Dysplasia (BPD). We propose to conduct a randomized trial of early (less than 3 days of age) treatment with intravenous azithromycin versus expectant management for VLBW infants with Ureaplasma spp. respiratory tract infection with the following specific aims: (1) Determine microbiological efficacy, pharmacokinetics, and safety of azithromycin treatment for eradication of Ureaplasma spp. in preterm infants, (2) Determine the respiratory outcomes of infants in the two treatment groups and those without respiratory tract Ureaplasma spp. infection

ELIGIBILITY:
Inclusion Criteria:

* Infants weighing <1250 grams at birth with respiratory distress syndrome who have respiratory infection with Ureaplasma sp organisms.

Exclusion Criteria:

* Severe respiratory distress syndrome with survival unlikely >7 days, Congenital malformations

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Schelonka, MD, Principal Investigator — University of Alabama at Birminham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Treatment With Azithromycin: Azithromycin (10mg/kg/day) start < 72 hours of age for 10 days
- Expectant (Usual) Management: Intervention at the discretion of the attending physician
Period: Overall Study
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Efficacy of Azithromycin Treatment for Eradication of Ureaplasma Spp. in Preterm Infants
Description: Number of subjects without ureaplasma spp at 100 days after study entry or at hospital discharge in subjects receiving therapy
Time Frame: 100 days or discharge from hospital
Population: Unable to determine efficacy due to low enrollment
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Respiratory Outcomes as Determined by Subjects Without Respiratory Tract Ureaplasma Spp Infection in Subjects in the Two Treatment Groups
Description: Absence of Ureaplasma spp infection is determined by the total number of days with positive pressure ventilation, (conventional ventilation or nasal continuous positive pressure) and oxygen therapy. The mean number of days was used to compare the two treatment groups.
Time Frame: from baseline to 100 days or discharge from Hospital, which ever comes first
Measure: Mean (Full Range); unit: days
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Number analyzed (Participants) | 5 | 2
days | 09.4 [0 to 23] | 2.5 [0 to 5]

3. Primary Outcome: Pharmacokinetics (PK) of Azithromycin Treatment for Eradication of Ureaplasma Spp. in Preterm Infants
Description: Pharmacokinetic measures (AUC12) of subjects receiving azithromycin who had eradication of ureaplasma spp.at either day 100 or discharge day which ever comes first.
Time Frame: 100 days or discharge from hospital
Population: Unable to determine Pharmacokinetics (PK) data due to low enrollment
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Safety of Azithromycin Treatment for Eradication of Ureaplasma Spp. in Preterm Infants
Description: Number of serious of adverse event experienced by subjects treated with azithromycin
Time Frame: from day 1 of study drug through 100 days or discharge from hospital, which ever comes first
Measure: Mean (Full Range); unit: number of events
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Number analyzed (Participants) | 5 | 2
number of events | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: enrollment through 100 days or discharge which ever is first
Arm/Group | Early Treatment With Azithromycin | Expectant (Usual) Management
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

LIMITATIONS AND CAVEATS:
Early termination due to small number enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No